CLINICAL TRIAL: NCT03564145
Title: A Multi-Center, Open-Label, Long-Term Safety Study of S5G4T-1 to Evaluate the Safety of S5G4T-1 in Papulopustular Rosacea Patients
Brief Title: A Long-Term Safety Study of S5G4T-1 in the Treatment of Papulopustular Rosacea
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Per protocol, the Sponsor could terminate the study once 300 participants completed a total of 28 weeks of treatment and 100 participants completed a total of 52 weeks.
Sponsor: Sol-Gel Technologies, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGT-54-07
Record Dates: First submitted 2018-06-10; First posted 2018-06-20 (Actual); Results first posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Papulopustular Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- S5G4T-1 (Experimental): Participants will topically apply S5G4T-1 cream, once daily to face for 40 weeks.
  Interventions: Drug: S5G4T-1

INTERVENTIONS:
Drug: S5G4T-1 — Once a day topical cream
  Other Names: Encapsulated Benzoyl Peroxide (E-BPO) Cream

SUMMARY:
To assess the safety of S5G4T-1 when applied once daily for up to 40 weeks in participants with papulopustular rosacea who completed either Study SGT-54-01 (NCT03448939) or Study SGT-54-02 (NCT03564119).

DETAILED DESCRIPTION:
This is a long-term safety study for participants who completed either study SGT-54-01 or SGT-54-02. Participants will be admitted into the study only after a written informed consent has been obtained and not missing more than 1 visit of Visits 3, 4 or 5 in these studies. Eligible participants for enrollment will apply the study product, S5G4T-1, daily for up to an additional 40 weeks for a total of up to 52 weeks for some participants.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must sign an Institutional Review Board (IRB) approved written informed consent for the extension study.
2. Participants must complete 12 weeks or within the Week 12 window time (± 4 days) of the double-blind treatment period of Study SGT-54-01 or Study SGT-54-02 and missed not more than 1 visit of Visits 3, 4 or 5 in Study SGT-54-01 or Study SGT-54-02.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 547 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2019-11-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sol-Gel, Rochester, New York, United States

REFERENCES:
- [Derived] Werschler WP, Sugarman J, Bhatia N, Baldwin H, Green LJ, Nov O, Ram V, Levy-Hacham O, Stein Gold L. Long-term Efficacy and Safety of Microencapsulated Benzoyl Peroxide Cream, 5%, in Rosacea: Results From an Extension of Two Phase III, Vehicle-controlled Trials. J Clin Aesthet Dermatol. 2023 Aug;16(8):27-33. PMID 37636251

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who completed either Study SGT-54-01 (NCT03448939) or Study SGT-54-02 (NCT03564119) were assigned to treatment with S5G4T-1 (Encapsulated Benzoyl Peroxide [E-BPO] cream).
Groups:
- S5G4T-1: Participants topically applied S5G4T-1 cream, once daily to face for 40 weeks.
Period: Overall Study
Arm/Group | S5G4T-1
Started | 547
Received at Least 1 Dose of Study Drug | 535
Completed | 323
Not Completed | 224
Not completed — Adverse Event | 4
Not completed — Lost to Follow-up | 21
Not completed — Protocol Violation | 2
Not completed — Withdrawal by Subject | 48
Not completed — Study Terminated by Sponsor | 146
Not completed — Physician Decision | 1
Not completed — Other Than Specified | 1
Not completed — Pregnancy | 1

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received at least 1 confirmed dose of S5G4T-1 and had at least 1 assessment.
Arm/Group | S5G4T-1
Number analyzed (Participants) | 535
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.5 (13.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 382
  Male | 153
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 155
  Not Hispanic or Latino | 380
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 36
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 1
  White | 492
  More than one race | 3
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE was defined as any untoward medical occurrence in a participant, which does not necessarily have a causal relationship with the study drug. Abnormalities presented at Baseline were considered AEs if they reoccurred after resolution or worsen during the AE collection period. An SAE was defined as any AE that, in the view of either the Investigator or Sponsor, resulted in any of the following outcomes as fatal, life-threatening, required hospitalization or prolongation of existing hospitalization, persistent or significant disability/incapacity, a congenital anomaly/birth defect, or an important medical event. A summary of all SAEs and Other AEs (non-serious) regardless of causality is located in 'Reported Adverse Events' Section.
Time Frame: Baseline up to Week 52
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | S5G4T-1
Number analyzed (Participants) | 535
Participants
  AEs | 185
  SAEs | 10

ADVERSE EVENTS:
Time Frame: Baseline (Day 0) through end of study (Week 52)
Description: The safety population included all participants who received at least 1 confirmed dose of S5G4T-1 and had at least 1 assessment.
Arm/Group | S5G4T-1
All-Cause Mortality (participants affected / at risk) | 0/535
Serious Adverse Events (participants affected / at risk) | 10/535
Other Adverse Events (participants affected / at risk) | 98/535
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | S5G4T-1 (N=535)
Arrhythmia (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Embolic stroke (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Mastectomy (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | S5G4T-1 (N=535)
Nasopharyngitis (Infections and infestations) | 29
Upper respiratory tract infection (Infections and infestations) | 12
Urinary tract infection (Infections and infestations) | 9
Influenza (Infections and infestations) | 8
Sinusitis (Infections and infestations) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 7
Application site erythema (General disorders) | 7
Application site pain (General disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Hypertension (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the Principal Investigator is not permitted to discuss or publish trial results without Sponsor approval.

DOCUMENTS (2):
  • Study Protocol (2018-11-27): https://cdn.clinicaltrials.gov/large-docs/45/NCT03564145/Prot_002.pdf
  • Statistical Analysis Plan (2019-11-18): https://cdn.clinicaltrials.gov/large-docs/45/NCT03564145/SAP_001.pdf